CLINICAL TRIAL: NCT06348368
Title: Refractive and Corneal Topographic Characteristics in Upper Egypt Children With High Cylinder
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Elshimaa A.Mateen, Clinical professor, Sohag University
Other Study IDs: Soh-Med-23-01-29
Record Dates: First submitted 2024-03-27; First posted 2024-04-04 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Corneal Ectasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 (control group): Children with normal Pentacam and with no refractive errors
  Interventions: Other: Pentacam and autorefractometry
- Group 2 (children with high cylinder and no corneal topographic abnormalities): Children with high cylinder without corneal topographic ectasia.
  Interventions: Other: Pentacam and autorefractometry
- Group 3 (Children with high cylinder and corneal ectatic changes).: Children with high cylinder and corneal ectatic changes
  Interventions: Other: Pentacam and autorefractometry

INTERVENTIONS:
Other: Pentacam and autorefractometry — Pentacam to detect corneal topographic changes. Auto-refractometry to assess refraction condition of the children

SUMMARY:
Refractive and Corneal Topographic Characteristics in upper Egypt children with high cylinder: A cross sectional study

DETAILED DESCRIPTION:
Astigmatism is defined as, a refractive condition in which refractive light fails to form a focus on the retina, it accounts for about 13% of refractive errors. It is frequent and correctable cause of visual impairment in children whether associated with spherical errors or not.

Astigmatism, is the refractive error of the highest clinical importance, being associated with reduced visual acuity with subsequent development of refractive amblyopia.

High cylinder in children belong to areas of hot and dry climates, makes exclusion of keratoconus is mandatory. Population in the African continent, the Mediterranean countries, Central and South America, and the Indian subcontinent usually have the habit of eye rubbing because of bothering symptoms of dryness, itching, atopy, allergy and vernal keratoconjunctivitis, which is the severe form of allergic conjunctivitis.

Eye rubbing causes thinning of keratocyte and increases the prevalence of keratoconus.

Keratoconus in children (diagnosed before the age of eighteenth) is less common but more aggressive than that of the adults, due to the dynamic nature of the young cornea. Few studies in the literature reported the prevalence and incidence of keratoconus in children.

Pentacam is an advanced instrument with a rotating Scheimpflug camera for scanning the anterior and posterior corneal surfaces. Its measurements of the corneal thickness and posterior elevation have been proved to be of high reproducibility and repeatability.

ELIGIBILITY:
Inclusion Criteria:

- Upper Egypt children with high cylinder(refractive errorr).

Exclusion Criteria:

* Children below age of 7 years old (uncooperative), patients above age of 18 years old.Patients with corneal scars

Ages: 7 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children live in upper Egypt with high cylinder and no corneal scar.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Values anterior and posterior corneal elevation values by pentacam. | one year
  Corneal topgraphic changes in children with high cylinder in upper Egypt

CONTACTS AND LOCATIONS:
Overall Officials: Elshimaa A.Mateen, Principal Investigator — Assistant professor of ophthalmology, Sohag University
Locations (1):
- Elshimaa A.Mateen, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided